CLINICAL TRIAL: NCT06596681
Title: A Study of the Safety and Tolerability of GA in the Treatment of Patients With Refractory Neuropathic Pain
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, chief physician, professor, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-157-03
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Pain, Intractable
Keywords: Refractory neuropathic pain; GA; clozapine; safety
MeSH Terms: conditions — Pain, Intractable; Neuralgia

STUDY DESIGN:
Intervention Model Description: A group of patients with refractory neuropathic pain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GA intracranial injection combined with oral clozapine (Experimental): Patients were first given intracranial injections of GA , followed by the oral clozapine.
  Interventions: Genetic: GA+clozapine

INTERVENTIONS:
Genetic: GA+clozapine — Patients were first given intracranial injections of GA and observed for 14-28 days, followed by a dose-climbing trial of clozapine medication, and finally, after the investigators had determined an effective dose of clozapine, the patients were given a fixed dose of clozapine orally for three months.

SUMMARY:
Previous studies have shown that the anterior cingulate cortex is involved in the regulation of pain and its associated negative emotions, that pyramidal neurons are highly excitable in chronic neuropathic pain conditions, and that silencing of pyramidal neurons can eliminate pain. The aim of this study was to evaluate the safety, tolerability, and efficacy of intracranial injection of GA (containing the hM4Di gene) in the anterior cingulate cortex in combination with oral clozapine for the treatment of refractory neuropathic pain.

DETAILED DESCRIPTION:
There is no effective treatment for refractory neuropathic pain, and this study aims to develop new treatments. Previous studies have shown that the anterior cingulate cortex is involved in the regulation of pain and its associated negative emotions, that pyramidal neurons are highly excitable in chronic neuropathic pain conditions, and that silencing of pyramidal neurons can eliminate pain. Animal studies have shown that inhibition of anterior cingulate cortex neurons using chemical genetics can effectively eliminate pain responses. Our team has obtained similar therapeutic effects with chemical genetics in mouse models of central pain, bone cancer pain, migraine, and nerve injury. In this study, a chemogenetic approach was used to express designer receptors exclusively activated by designer drug (hM4Di) in the anterior cingulate cortex, which binds to clozapine to inhibit neuronal excitability. The aim of this study was to evaluate the safety, tolerability, and efficacy of intracranial injection of GA (containing the hM4Di gene) in the anterior cingulate cortex in combination with oral clozapine for the treatment of refractory neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a definitive diagnosis of neuropathic pain, including but not limited to painful diabetic peripheral neuropathy, trigeminal neuralgia, and post-stroke pain, aged 18-65 years old (regardless of gender), with:

   1. Regularised treatment with conventional medical therapy (including, but not limited to, medication, physiotherapy, cognitive therapy, nerve blocks and other non-invasive or minimally invasive treatments) for at least 3 months with no symptomatic relief or emergence of tolerance, as assessed by the investigator
   2. Pharmacological treatment means a full course of treatment with at least two first-line medications, as assessed by the investigator
2. Mean visual analogue scale (VAS) value ≥4 cm and/or mean numerical rating scale (NRS) value ≥4 points within one week of baseline at enrolment
3. Subjects who have had a stable analgesic regimen for at least 30 days prior to the intensity of pain described in Inclusion Criterion 2 and agree not to arbitrarily change the type and dose of medication that they are currently taking until the end of the period of assessment of the effectiveness of this trial, as assessed by the investigator
4. Subjects volunteered to participate in the trial and gave fully informed consent to sign an informed consent form
5. Have stable neurological status as assessed by the researcher through motor, sensory and reflex functions
6. Subjects are considered reliable and able to comply with the trial protocol (e.g., able to understand and complete relevant scales), visit protocols, and medication administration, according to the investigator's judgement
7. Subjects of childbearing potential agree to sign an informed consent form and have no plans to have children during the study period and voluntarily use effective contraception (oral contraceptives are prohibited) and do not plan to donate sperm or eggs

Exclusion Criteria:

* 1.In patients with painful diabetic peripheral neuropathy, amputation due to diabetes mellitus or large (≥3cm) and/or gangrenous ulcers on the lower limbs 2.Currently diagnosed with progressive neurological disorders such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, tumours of the brain or spinal cord, and neurodegenerative disorders, as determined by the investigators 3.Have a chronic systemic disease that, as assessed by the investigator, may affect the subject's participation in the study, including but not limited to:

  1. suffering from severe cardiopulmonary disease such as unstable angina, myocardial infarction, severe arrhythmia, recurrent asthma attacks, etc;
  2. Malignant tumours of the central nervous system or other systems. 4.Current status such as coagulation disorders, bleeding tendencies, platelet dysfunction, severely reduced function due to underlying cardiac/pulmonary disease, progressive peripheral vascular disease, or poorly controlled diabetes mellitus, and subjects who may be suffering from a relevant disease state that affects surgery as assessed by the investigator 5.Currently on anticoagulants and unable to stop them 6.Localised infection or active systemic infection at the anticipated surgical access site 7.History of previous intracranial surgical treatment (except for minimally invasive paracentesis for diagnostic tests, etc.) 8.Patients with severe psychiatric symptoms (e.g., major depression, schizophrenia, etc.) or significant suicidal tendencies or assessed by the investigator to be unable to complete the clinical trial 9. Pre-existing or concomitant severe hepatic dysfunction, renal dysfunction, cardiac dysfunction (in which severe hepatic dysfunction is defined as ALT ≥ 2.0 times the upper limit of normal or AST ≥ 2.0 times the upper limit of normal; severe renal dysfunction refers to a CRE ≥ 1.5 times the upper limit of normal or an eGFR < 40mL/min/1.73m2; and severe cardiac dysfunction refers to an NYHA score of grade 3-4) ，delirium, hypotension, epilepsy, glaucoma, myelosuppression or leukopenia, severe central nervous system depression, or coma from any cause 10. Subjects with abnormal laboratory test values:

  <!-- -->

  1. white blood cell count <3.5 x 109/L and neutrophil count <1.0 x 109/L
  2. Platelet (PLT) <75 x 109/L
  3. Coagulation: prothrombin time and activated partial thromboplastin time >1.5 x ULN
  4. Blood adeno-associated virus (AAV) antibody titre >1:1000 11.Patients taking drugs that cause granulocyte deficiency or have myelosuppressive effects 12.Patients with granulocyte deficiency or severe granulocytopenia due to prior clozapine use 13.Patients with contraindications and/or allergies to medications during the trial (e.g. clozapine or other components of clozapine, contrast agents, etc.) 14.Have gastrointestinal diseases (Crohn's disease, acute or chronic pancreatitis, paralytic intestinal obstruction, etc.) or major gastrointestinal surgeries that affect the absorption, metabolism and excretion of drugs, etc.

     15.Subjects had received any gene or cellular therapy 16. Known history of alcohol, drug abuse 17.Patients participating in other clinical trials or applying other investigational biologics, drugs or devices within six months prior to screening 18.Contraindications to MRI and functional MRI (e.g. claustrophobia, metallic foreign bodies in the body) 19.Clozapine-related serious adverse reactions are considered a screening failure if they occur during the screening period, at the judgement of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE)/serious adverse events (SAE) as assessed by CTCAE v5.0 | up to 28 weeks
  Patient-Reported Adverse Events, Abnormalities on Physical Examination, and Abnormalities in Laboratory Tests

SECONDARY OUTCOMES:
effectiveness: the degree of pain improvement was assessed by visual analogue scale (VAS). | Weeks 4, 8, and 12 of the effectiveness observation period
  The degree of pain improvement was assessed by visual analogue scale (VAS). VAS Score: i.e. Pain Scale Rating, which assesses the severity of pain using visual analogue methods. The scale uses a 10cm long straight line with '0' cm and '10' cm at each end, with 0 indicating no pain and 10 indicating unbearable severe pain.
effectiveness: the pain improvement was assessed by Brief pain inventory (BPI) scale. | Weeks 4, 8, and 12 of the effectiveness observation period
  the pain improvement was assessed by Brief pain inventory (BPI) scale. BPI: Evaluates pain severity and functional interference. Part 1 (Severity): Current pain, average pain (24h), worst pain (24h), least pain (24h), pain relief from treatments. Part 2 (Interference): Impact on general activity, mood, walking ability, work, relationships, sleep, and enjoyment of life.
effectiveness: the degree of sleep quality improvement was assessed by Insomnia Severity Index (ISI). | Weeks 4, 8, and 12 of the effectiveness observation period
  The degree of sleep quality improvement was assessed by Insomnia Severity Index (ISI). ISI scale: 7 entries, each rated 0-4. The total score ranges from 0-28, and the higher the score the greater the severity of insomnia.
effectiveness: the sleep quality improvement was assessed by Daily Sleep Interference Scale (DSIS). | Up to 28 weeks
  the sleep quality improvement was assessed by Daily Sleep Interference Scale (DSIS). DSIS: An 11-point Likert scale ranging from 0 ("Pain did not interfere with sleep") to 10 ("Pain completely interfered with sleep" [inability to sleep due to pain]). Subjects will recall sleep interference over the preceding 24 hours each morning and record scores.
effectiveness: the depression improvement was assessed by Hamilton depression (HAMD) scale. | Weeks 4, 8, and 12 of the effectiveness observation period
  The depression improvement was assessed by Hamilton depression (HAMD) scale. HAMD: 17-item version implemented in this protocol. Trained raters will conduct combined evaluations through structured interviews and behavioral observations.
effectiveness: the degree of depression improvement was assessed by Patient Health Questionnaire-9 (PHQ-9). | Weeks 4, 8, and 12 of the effectiveness observation period
  The degree of depression improvement was assessed by Patient Health Questionnaire-9 (PHQ-9).PHQ-9: Used to screen patients for depressive disorders. The PHQ-9 scale has 9 items, each of which is a 4-point scale from 0-3. According to the scale, the PHQ-9 score is divided into 5 groups: 0-4, 5-9, 10-14, 15-19, and 20-27, corresponding to no, mild, moderate, moderately severe, and severe depression, respectively.
effectiveness: the anxiety improvement was assessed by Hamilton anxiety (HAMA) scale. | Weeks 4, 8, and 12 of the effectiveness observation period
  The anxiety improvement was assessed by Hamilton anxiety (HAMA) scale. HAMA: 14-item clinician-administered scale recognized as a primary diagnostic tool for anxiety disorders according to the Chinese Classification of Mental Disorders-3 (CCMD-3).
effectiveness: the degree of anxiety improvement was assessed by Generalized Anxiexy Disorde-7 (GAD-9). | Weeks 4, 8, and 12 of the effectiveness observation period
  The degree of anxiety improvement was assessed by Generalized Anxiexy Disorde-7 (GAD-9). The GAD-7 is a widely used self-assessment scale for anxiety symptoms that has been used in recent years to screen not only for anxiety disorders, but also for panic disorder, social anxiety disorder, and post-traumatic stress disorder. The scale consists of 7 items that rate tension, uncontrollable worry, excessive worry, inability to relax, inability to sit still, irritability, and feelings of foreboding. The number of days in the last 2 weeks that the target symptom was present was assessed: 0 for no symptoms, 1 for a few days, 2 for more than half of the days, and 3 for almost every day. A total score of 5 to 9 is considered mild, 10 to 14 is moderate, and 15 to 21 is severe.
effectiveness: the degree of quality of life improvement was assessed by EuroQOL, 5 Domains, 5 Levels (EQ-5D-5L). | Weeks 4, 8, and 12 of the effectiveness observation period
  The degree of quality of life improvement was assessed by EuroQOL, 5 Domains, 5 Levels (EQ-5D-5L). The EQ-5D-5L is a set of standardised scales to measure health status. The EQ-5D-5L consists of two parts, the EQ-5D-5L Health Descriptor System and the EQ-VAS. The EQ-5D-5L Health Descriptor System describes five dimensions: mobility, Self-Care, Usual Activities, Pain/Comfort, Anxiety/Depression. Each dimension consists of five levels: 1 No difficulty, 2 Some difficulty, 3 Moderate difficulty, 4 Severe difficulty, and 5 Unable to perform/very severe difficulty. Responses to the five dimensions generate a five-digit code describing the state of health, with a state of health of 11111 indicating no problems on any of the five dimensions.The EQ-VAS records the self-assessed state of health on a vertical, visually analogue scale, with the ends of the scale labelled 'the best health you can imagine' and 'the worst health you can imagine'.
effectiveness: the quality of life improvement was assessed by Patient global impression of change (PGIC). | Weeks 4, 8, and 12 of the effectiveness observation period
  the quality of life improvement was assessed by Patient global impression of change (PGIC). PGIC: A 7-point scale assessing subjects' overall perception changes following treatment: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse.
immunogenicity endpoint: AAV antibody titres | up to 28 weeks
  Use of specific antibodies for AAV antibody titre testing
Antigen-specific T-cell responses | Up to 28 weeks
  Antigen-specific T-cell responses
Pharmacokinetic profile: Carrier genome levels in urine, blood, tears, nasal secretions | up to 28 weeks
  Carrier genome levels in urine, blood, tears, nasal secretions

OTHER OUTCOMES:
fMRI: Neuronal activation in ACC brain regions and connectivity of ACC brain regions with other brain regions | up to 28 weeks
  fMRI: is a radiation-free, non-invasive functional imaging technique that detects the level of neuronal activation in brain tissue by probing blood oxygen saturation and water levels in brain tissue. In this programme, local brain activity (activation of neurons in brain regions) and brain integration (functional connectivity between brain regions) are assessed, especially in the ACC brain region.
Drug Dose Reduction | up to 28 weeks
  After the patient is treated with GA intracranial injections combined with oral clozapine and the pain symptoms improve, the previous analgesic medication of patients may be considered to be gradually tapered off

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, Doctor, Study Chair — Beijng tiantan hospital; Hua Pan, Doctor, Study Director — Beijng tiantan hospital; Fang Luo, Doctor, Study Director — Beijng tiantan hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No